CLINICAL TRIAL: NCT03198182
Title: A Randomized, Parallel, Placebo-Controlled, Multiple Dose Study to Evaluate the Safety to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of BMS-986036 in Healthy Japanese and Non-Japanese Subjects
Brief Title: A Study to Test the Effects of BMS-986036 on the Body in Healthy Japanese and Non-Japanese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: MB130-057
Record Dates: First submitted 2017-06-22; First posted 2017-06-26 (Actual); Last update posted 2019-05-01 (Actual); Status verified 2019-04

CONDITIONS: Metabolics
MeSH Terms: interventions — Pegbelfermin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Module A (Experimental): BMS-986036 Arm
  Interventions: Drug: BMS-986036
- Module B (Placebo Comparator): Placebo Arm
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Specified dose on specified days
  Arms: Module B
Drug: BMS-986036 — Specified dose on specified days
  Arms: Module A

SUMMARY:
The purpose of this study is to evaluate safety, and tolerability of BMS-986036 and the effects the drug has on the body

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects, as determined by no clinically significant deviations from normal in medical history, physical examination, electrocardiograms (ECGs), and clinical laboratory determinations
* Body mass index (BMI) of 25 to 40 kilogram / square meter (kg/m2), inclusive
* Additional criterion for Japanese subjects: Subjects must be first generation Japanese (born in Japan and not living outside of Japan for > 10 years, and both parents are ethnically Japanese)

Exclusion Criteria

* Presence of any factors that would predispose the subject to infection (extensive periodontal disease that warrants surgical or medical treatment, unhealed open wounds)
* Any bone trauma (fracture) or bone surgery (hardware placement, joint replacement, bone grafting, or amputation) within 3 months of study drug administration
* Known or suspected autoimmune disorder, excluding vitiligo

Other protocol defined inclusion/exclusion criteria could apply

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 63 (Actual)
Dates: Start 2017-06-28 (Actual); Primary Completion 2017-09-22 (Actual); Study Completion 2017-09-22 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) | Up to 42 days
  Safety
Incidence of serious adverse events (SAEs) | Up to 42 days
  Safety

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- WCCT Global, Cypress, California, United States

REFERENCES:
- See also: BMS Clinical Trial Patient Recruiting — http://bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry Form — http://www.bms.com/clinical_trials/Pages/Investigator_inquiry_form.aspx